CLINICAL TRIAL: NCT05730153
Title: Clinical and Radiographic Evaluation of Advanced Platelet Rich Fibrin and Open Debridement in Management of Periodontal Suprabony Defects
Brief Title: Advanced Platelet-rich Fibrin Combined With Open Debridement in Management of Suprabony Periodontal Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Naglaa Elwakeel, professor, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMD 3-22
Record Dates: First submitted 2023-02-07; First posted 2023-02-15 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-02

CONDITIONS: Periodontitis, Adult
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator)
  Interventions: Biological: advanced PRF
- group 2 (Sham Comparator)
  Interventions: Biological: advanced PRF

INTERVENTIONS:
Biological: advanced PRF — advanced PRF+ surgery

SUMMARY:
in this clinical trial, patients with periodontal defects will be treated with advanced platelet-rich fibrin in conjunction with open debridement

DETAILED DESCRIPTION:
two groups of patients with suprabony defects, one will be treated with advanced platelet-rich fibrin in conjunction with open debridement and the other will be treated with open debridement alone. subjects will be evaluated for evidence of bone formation after 6 months of therapy

ELIGIBILITY:
Inclusion Criteria:

* patients with periodontal suprabony defects.

Exclusion Criteria:

* pregnant females.
* smokers.
* systemic disease that contraindicate surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
clinical evaluation | 6 months
  Rate of probing pocket depth reduction

SECONDARY OUTCOMES:
radiographic evaluation | 6 months
  Rate of bone formation by digital radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Faculty of Dentistry, Cairo, Egypt